CLINICAL TRIAL: NCT04924231
Title: Effect of 1.8-mm Steep-axis Clear Corneal Incision on the Posterior Corneal Astigmatism in Candidates for Toric IOL Implantation
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-407
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: astigmatism — astigamatism at least 1 month after the cataract surgery

SUMMARY:
we aimed to analyze the effects of cataract surgery using a 1.8-mm steep-axis clear corneal incision (CCI) on the posterior corneal surfaces based on the keratometry from the rotating Scheimpflug imaging device (Pentacam HR) in candidates for toric intraocular lens (IOL) implantation

DETAILED DESCRIPTION:
Preoperative and at least 1-month postoperative data measured by Pentacam HR were collected in patients for toric IOL implantation. Surgically induced astigmatism on the posterior cornea (P-SIA) was calculated based on the preoperative and postoperative keratometric data, and the related factors of P-SIA were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged at least 45 years old who were scheduled for cataract surgery; (2) regular corneal astigmatism ≥ 1.0 D; (3) the imaging quality parameter (QS) of Pentacam HR was "OK"; and (4) follow-up time ≥1.0 month.

Exclusion Criteria:(1) irregular corneal astigmatism; (2) corneal scar, corneal degeneration, pterygium invading the optic zone; (3) corneal endothelium count<1,000/mm2, corneal endothelial dystrophy, iritis, glaucoma and retinal disease; (4) history of eye surgery, such as corneal refractive surgery, corneal transplantation and retinal surgery; (5) the main incision was expanded or sutures were used during surgery; and (6) some postoperative complications, such as persistent corneal edema, Descemet's membrane detachment and poor wound healing, and any others that might affect the measurement results of the Pentacam HR during the follow-up period.

-

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients, who underwent cataract surgery with a 1.8-mm steep-axis CCI at the Eye Center, the Second Affiliated Hospital of Zhejiang University
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
corneal astigmatism | post 1 month
  postoperative anterior, posterior and total corneal astigmatism

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided